CLINICAL TRIAL: NCT04092543
Title: Prediction of Outcome After Acute Stroke: Validation of CT-DRAGON Versus a Simplified CT-DRAGON Score
Brief Title: Validation of DRAGON Versus a Simplified DRAGON/Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, Principal Investigator, Ziekenhuis Oost-Limburg
Other Study IDs: DRAGON
Record Dates: First submitted 2019-08-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Stroke, Acute
Keywords: CT-DRAGON score
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: All patients diagnosed with a stroke are collected in the database.

SUMMARY:
The CT-DRAGON score can predict long-term functional outcome after acute stroke treated by thrombolysis. However, implementation in clinical practice is hampered by a lack of validation in the broad spectrum of stroke patients undergoing thrombectomy, whether or not in combination with thrombolysis or conservative treatment. Furthermore, the CT-DRAGON score considers multiple items, which are not always readily available in every setting. This study aims to investigate whether either a simplified version of the CT-DRAGON score with only three clinical items or a machine learning technique could be as powerful and more feasible.

DETAILED DESCRIPTION:
The investigators aim to validate the CT-DRAGON score in all ischaemic stroke localisations and for all treatment options, including a conservative treatment policy. The predictability will then be compared with on the one hand simplified prognostic models that include only a selective set of highly predictive parameters that have already been described in the literature, such as patient age, National Institutes of Health Stroke Scale (NIHSS) and pre-stroke modified Rankin Scale (mRS). On the other hand, machine learning techniques, that incorporate a large set of variables and have recently shown some promising results, will also be applied to predict long-term outcome after ischaemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with a stroke

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with a stroke will be analyzed in the database starting from March 1, 2019 until August 1 2021
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale at day 90 | 90 days after the onset of stroke
  The modified rankin scale will be assessed at 90 days at a consultation or by a telephonic interview which is standard of care in the hospital. The scale runs from 0-6, running from perfect health without symptoms to death.
Modified Rankin Scale at 7 days after discharge | 7 days after discharge at the hospital
  The modified rankin scale will be assessed at 7 days after discharge by a telephonic interview which is standard of care in the hospital. he scale runs from 0-6, running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
PROMIS 10 questionnaire at 7 days after discharge | 7 days after discharge
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a publically available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life.The scoring system of the PROMIS Global-10 allows each of the individual items to be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health.The summed total is reported as 0 to 48 with higher scores reflecting less pain and better function.
PROMIS 10 questionnaire at 90 days after the onset of stroke | 90 days after the onset of stroke
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a publically available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life.The scoring system of the PROMIS Global-10 allows each of the individual items to be examined separately to provide specific information about perceptions of physical function, pain, fatigue, emotional distress, social health and general perceptions of health. The summed total is reported as 0 to 48 with higher scores reflecting less pain and better function.
NIHSS at 90 days after the onset of stroke | 90 days after the onset of stroke
  Change in NIHSS over time: baseline (diagnosis stroke), 3 months and one year follow-up. The National Institutes of Health Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Analysis of the hospitalization cost after the onset of stroke | 90 days after the onset of stroke
  90 days after the onset of stroke, all hospitalization costs will be analyzed per patient. All costs related to stroke in our hospital will be analyzed (surgery, clinical investigations, revalidation therapy etc) by our financial department.

CONTACTS AND LOCATIONS:
Overall Officials: dieter Mesotten, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lesenne A, Grieten J, Ernon L, Wibail A, Stockx L, Wouters PF, Dreesen L, Vandermeulen E, Van Boxstael S, Vanelderen P, Van Poucke S, Vundelinckx J, Van Cauter S, Mesotten D. Prediction of Functional Outcome After Acute Ischemic Stroke: Comparison of the CT-DRAGON Score and a Reduced Features Set. Front Neurol. 2020 Jul 31;11:718. doi: 10.3389/fneur.2020.00718. eCollection 2020. PMID 32849196